CLINICAL TRIAL: NCT03148691
Title: A Phase 2 Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Study of the Safety and Effectiveness of A-101(Hydrogen Peroxide) Topical Solution in Subjects With Seborrheic Keratosis Lesions on the Trunk, Extremities, and Face
Brief Title: A Randomized, Vehicle-Controlled Study of 2 Concentrations of A-101 for the Treatment of Seborrheic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-101-SEBK-204
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Seborrheic Keratosis
MeSH Terms: conditions — Keratosis, Seborrheic | interventions — N-phenylacetoaminomethylene-DL-p-nitrophenylalanine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vehicle (Placebo Comparator): Vehicle Topical Solution
  Interventions: Drug: A-101
- A-101 Low Dose (Active Comparator): A-101 Low Dose Topical Solution
  Interventions: Drug: A-101
- A-101 High Dose (Active Comparator): A-101 High DoseTopical Solution
  Interventions: Drug: A-101

INTERVENTIONS:
Drug: A-101 — Topical Solution

SUMMARY:
The primary objective of this study is to evaluate the safety and effectiveness of 2 concentrations of A-101 compared to Vehicle for the treatment of 4 seborrheic keratosis (SK) Target Lesions on the trunk, extremities and face.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and effectiveness of 2 concentrations of A-101 compared to Vehicle for the treatment of 4 seborrheic keratosis (SK) Target Lesions on the trunk, extremities and face.

The secondary objectives of this study include duration of response of A-101. During the study, the investigator will identify 4 eligible SK Target Lesions on each subject on the trunk, extremities and face. For each subject, at least 1 SK Target Lesion must be on the face and at least 1 Target Lesion must be on the trunk or extremities. The Target Lesions will be treated at a maximum of two treatment visits.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to comprehend and is willing to sign an informed consent for participation in this study.
2. Male or female ≥ 18 years old.
3. Subject has a clinical diagnosis of stable clinically typical seborrheic keratosis.
4. Subject has 4 appropriate seborrheic keratosis Target Lesions on the trunk, extremities and face, with at least 1 Target Lesion on the face and at least 1 Target Lesion on the trunk or extremities. The 4 identified Target Lesions must meet the requirements as defined below:

   1. Have a clinically typical appearance
   2. Have a Physician's Lesion Assessment of ≥ 2
   3. Length that is ≥ 5mm and ≤ 15mm
   4. Width that is ≥ 5mm and ≤ 15 mm
   5. Thickness that is ≤ 2mm
   6. Be a discrete lesion
   7. Be the only SK lesion present when centered in the area outlined by the provided circular template
   8. Not be covered with hair which, the in the investigator's opinion, would interfere with the study medication treatment or the study evaluations
   9. Not be in the intertriginous fold
   10. Not be on the eyelids
   11. Not be within 5mm of the orbital rim
   12. Not be pedunculated
5. Subject chemistry and complete blood count results are within normal limits. If any of the laboratory values are outside normal range, the treating investigator must assess the value/s as NOT clinically significant and document this in the subject's medical chart in order for the subject to be eligible for randomization.
6. Woman of childbearing potential must have a negative urine pregnancy test within 14 days of the first application of study drug and agree to use an active method of birth control for the duration of the study.
7. Subject is non-pregnant and non-lactating.
8. Subject is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair the evaluation of any Target Lesion or which exposes the subject to an unacceptable risk by study participation.
9. Subject is willing and able to follow all study instructions and to attend all study visits.

Exclusion Criteria:

1. Subject has clinically atypical and /or rapidly growing seborrheic keratosis lesions.
2. Subject has presence of multiple eruptive seborrheic keratosis lesions (Sign of Leser - Trelat).
3. Subject has current systemic malignancy.
4. Subject has used any of the following systemic therapies within the specified period prior to Visit 1:

   * Retinoids; 180 days
   * Corticosteroids; 28 days
   * Anti-metabolites (e.g., methotrexate); 28 days
5. Subject has used any of the following topical therapies within the specified period prior to Visit 1 on, or in a proximity to any Target Lesion, that in the investigator's opinion interferes with the study medication treatment or the study assessments:

   * LASER, light or other energy based therapy (e.g., intense pulsed light, photo-dynamic therapy; 180 days
   * Liquid nitrogen, electrodesiccation, curettage, imiquimod, 5-Fluorouracil, or ingenol mebutate; 60 days
   * Hydrogen peroxide: 90 days
   * Retinoids; 28 days
   * Microdermabrasion or superficial chemical peels; 14 days
   * Corticosteroids or antibiotics; 14 days
6. Subject would require the use of any topical treatment (e.g. moisturizers, sunscreen) to any of the Target Lesions 12 hours prior to any study visit.
7. Subject currently has or has had any of the following within the specified period prior to Visit 1 on or in a proximity to any Target Lesion that, in the investigator's opinion, interferes with the study medication treatment or the study assessments:

   * Cutaneous malignancy; 180 days
   * Sunburn; currently
   * Pre-malignancy (e.g. actinic keratosis); currently
   * Body art (e.g. tattoos, piercing, etc.); currently
   * Excessive tan; currently. The use of self-tanning lotions/sprays are prohibited.
8. Subject has a history of sensitivity to any of the ingredients in the study medications.
9. Subject has any current skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage), or condition (e.g., sunburn, excessive hair, open wounds) that, in the opinion of the investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations.
10. Participation in another therapeutic investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Shanler, MD, Study Director — Aclaris Therapeutics, Inc.
Locations (9):
- United States (9):
  - Center for Dermatology and Dermatologic Surgery, Washington D.C., District of Columbia
  - Baumann Research Institute, Miami, Florida
  - MedaPhase, Inc, Newnan, Georgia
  - Union Square Laser Dermatology, New York, New York
  - Philadelphia Institute - Dermatology, Fort Washington, Pennsylvania
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Greenville Dermatology, Greenville, South Carolina
  - The Skin Wellness Center, PC Clinical Research Division, Knoxville, Tennessee
  - DermResearch Inc, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle | A-101 Low Dose | A-101 High Dose
Started | 50 | 103 | 100
Completed | 47 | 101 | 92
Not Completed | 3 | 2 | 8
Not completed — Protocol Violation | 1 | 2 | 7
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Other | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | A-101 Low Dose | A-101 High Dose | Total
Number analyzed (Participants) | 50 | 103 | 100 | 253
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 30 | 21 | 65
  >=65 years | 36 | 73 | 79 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (8.27) | 69.1 (8.75) | 70.0 (8.12) | 69.5 (8.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 59 | 67 | 157
  Male | 19 | 44 | 33 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 4 | 16
  Not Hispanic or Latino | 43 | 89 | 88 | 220
  Unknown or Not Reported | 4 | 5 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 8 | 16
  White | 46 | 98 | 92 | 236
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 103 | 100 | 253

OUTCOME MEASURES:

1. Primary Outcome: Mean of Per Subject Percentages of Target Lesions Judged to be Clear (PWA=0) at Visit 8
Description: Mean of per subject percentages of target lesions judged to be clear (PWA=0) at Visit 8
  Grade Descriptor
  0 Clear: no visible seborrheic keratosis lesion
  1. Near Clear: a visible seborrheic keratosis lesion with a surface appearance different from the surrounding skin (not elevated)
  2. Thin: a visible seborrheic keratosis lesion (thickness ≤ 1 mm)
  3. Thick: a visible seborrheic keratosis lesion (thickness > 1 mm)
Time Frame: Day 106
Measure: Mean (Standard Deviation); unit: Per-Subject Percent of Lesions Clear
Units Other Than Participants: Lesions
Arm/Group | Vehicle | A-101 Low Dose | A-101 High Dose
Number analyzed (Participants) | 47 | 101 | 92
Number analyzed (Lesions) | 188 | 404 | 368
Per-Subject Percent of Lesions Clear | 3.72 (10.4) | 49.5 (36.74) | 57.88 (35.92)

ADVERSE EVENTS:
Time Frame: 11.5 months; Treatment-emergent adverse events (TEAEs) had a start date on or after the date of Visit 2 (study day 1) and treatment-emergent serious adverse events had a start date on or after the date of Visit 1 (Screening). Collection continued through the subject's last visit or the end of the study, visit 8 (Day 106.)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation subject administered a study medication(s) and that did not necessarily have a causal relationship with the study medication.
  Safety summaries by study medication group will include listings by study medication of adverse events incidences within each MedDRA System Organ Class, and changes from pre-application values in vital signs.
Arm/Group | Vehicle | A-101 Low Dose | A-101 High Dose
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/103 | 0/100
Serious Adverse Events (participants affected / at risk) | 1/50 | 2/103 | 1/100
Other Adverse Events (participants affected / at risk) | 11/50 | 18/103 | 26/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=50) | A-101 Low Dose (N=103) | A-101 High Dose (N=100)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Syncope and Collapse (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=50) | A-101 Low Dose (N=103) | A-101 High Dose (N=100)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bundle Branch Block Left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid Oedema (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Ocular Hypertension (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bile Duct Obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Body Tinea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Post operative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood osmolarity decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT03148691/Prot_SAP_000.pdf